CLINICAL TRIAL: NCT04359251
Title: Avoiding High PEEP in COVID-19 Induced ARDS: a Multi-center Study
Brief Title: Different PEEP Settings of COVID-19 Induced ARDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Chun Pan, Dr, Southeast University, China
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: COVID-19 PEEP titration
Record Dates: First submitted 2020-04-13; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: COVID-19; Mechanical Ventilation Pressure High; Acute Respiratory Distress Syndrome
Keywords: ARDS; COVID-19; mechanical ventilation; PEEP
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Optimizing oxygenation (Experimental): Best oxygenation during PEEP titration
  Interventions: Other: Gas exchanges at different PEEP
- Optimizing compliance (Experimental): Best compliance during PEEP titration
  Interventions: Other: lung mechanics at different PEEP
- ARDSnet (Experimental): PEEP settings according to ARDSnet table
  Interventions: Other: Hemodynamics changes at different PEEP

INTERVENTIONS:
Other: Gas exchanges at different PEEP — Gas exchanges measurement at different PEEP
  Arms: Optimizing oxygenation
Other: lung mechanics at different PEEP — lung mechanics measurement at different PEEP
  Arms: Optimizing compliance
Other: Hemodynamics changes at different PEEP — Hemodynamics changes measurement at different PEEP
  Arms: ARDSnet

SUMMARY:
This was a multi-center prospective study. All consecutive severe cases of COVID-19 whose PO2/FiO2<300mmHg with invasive ventilation admitted to 5 fixed-point receive COVID-19 patients hospitals in Wuhan from 5 March to 15 March 2020 were included. Epidemiological, clinical data, lung mechanics, artery blood gas test and hemodynamics at three methods to titrate PEEP, optimizing oxygenation, optimizing compliance, ARDSnet. The study was approved by the Ethics Committee of Zhongda Hsopital, Southeast University.

DETAILED DESCRIPTION:
After PEEP titration, PEEP settings could be set by optimizing oxygenation, optimizing compliance, ARDSnet.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 patients with mechanical ventilation
* PO2/FIO2<300mmHg
* ages>18 years

Exclusion Criteria:

* pneumothorax
* pregnant
* hemodynamics is unstable

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Respiratory system compliance improvement | 20 minutes
  the respiratory system compliance was compared among three groups

SECONDARY OUTCOMES:
Gas echanges improvement | 20 minutes
  P/Fwere compared among three groups

OTHER OUTCOMES:
hemodynamics improvement | 20 minutes
  MAP were compared among three groups

CONTACTS AND LOCATIONS:
Overall Officials: Chun C Pan, Study Director — Zhongda hospital, Southeast University, Jiangsu, China
Locations (1):
- Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pan C, Lu C, She X, Ren H, Wei H, Xu L, Huang Y, Xia J, Yu Y, Chen L, Du B, Qiu H. Evaluation of Positive End-Expiratory Pressure Strategies in Patients With Coronavirus Disease 2019-Induced Acute Respiratory Distress Syndrome. Front Med (Lausanne). 2021 Jul 20;8:637747. doi: 10.3389/fmed.2021.637747. eCollection 2021. PMID 34355001